CLINICAL TRIAL: NCT05981430
Title: Fecal Microbiota Transplantation for Decolonization of Carbapenem-resistant Enterobacteriaceae: a Double Blind Randomized Controlled Trial
Brief Title: Fecal Microbiota Transplantation for Decolonization of Carbapenem-resistant Enterobacteriaceae
Acronym: FMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Ka Shing, Clinical assistant professor. https://medic.hku.hk/en/Staff/University-Academic-Staff/Dr-CHEUNG-Ka-Shing-Michael/Dr-CHEUNG-Ka-Shing-Michael-Profile, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 19-512
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection; Fecal Microbiota Transplantation
Keywords: FMT; CRE
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal microbiota transplant (Active Comparator): This group's subject will receive an infusion of 125mL fecal suspension via enema.
  Interventions: Biological: Fecal microbiota transplant
- Sham fecal microbiota transplant (Placebo Comparator): This group's subject will receive 125mL placebo enema comprised of normal saline with 15% glycerol and brown food colouring 204 (Americolorcorp) as a sham procedure.
  Interventions: Biological: Sham fecal microbiota transplant

INTERVENTIONS:
Biological: Fecal microbiota transplant — Active comparator will receive infusion of 125mL fecal suspension via enema
  Arms: Fecal microbiota transplant
Biological: Sham fecal microbiota transplant — Placebo comparator will receive 125mL placebo enema comprised of normal saline with 15% glycerol and brown food coloring 204 (Americolorcorp).
  Arms: Sham fecal microbiota transplant

SUMMARY:
The emergence of multidrug-resistant organisms (MDROs) has become one of the major threats to the healthcare system in Hong Kong in recent years. The situation is particularly worrisome for carbapenem-resistant Enterobacteriaceae (CRE). Taking Queen Mary Hospital as an example, the number of CRE cases has surged from 24 in year 2014 to 625 in year 2021. The case burden in Hong Kong is therefore substantial when all 43 public hospitals and institutions in Hong Kong are considered. With the widespread use of broad-spectrum antibiotics and active case screening, the number of CRE cases is expected to further increase in an exponential manner.

Given that colonization with MDROs is due to gut dysbiosis from antibiotic use, a normal intestinal microbiota is apparently crucial in protecting hosts from colonization with MDROs including CRE. Fecal microbiota transplantation (FMT), which involves the infusion of stool from a healthy donor to the gastrointestinal (GI) tract of a recipient, has gained popularity in recent years to restore colonic microbial diversity in various diseases associated with gut dysbiosis, e.g. Clostridium difficile (CD) infection, ulcerative colitis and even metabolic diseases. The investigators aim to conduct a double-blind randomized controlled trial to evaluate the benefit of FMT via lower GI delivery (enema) on CRE clearance.

DETAILED DESCRIPTION:
CRE colonization is associated with a 16.5% risk of infection with a 10% mortality rate. CRE also poses a tremendous strain on the healthcare cost as well as the medical/nursing manpower. The hospital stay is lengthened by two-fold for CRE-infected cases compared with non-infected cases. CRE carriers frequently have to stay in acute hospitals for extended periods of time after settling their acute illnesses, both because of the logistic infeasibility of them being transferred to rehabilitation units or nursing homes, which are devoid of isolation rooms.

Proactive measures have been implemented in hospitals worldwide to prevent the spread of MDROs, especially to vulnerable individuals. Such measures usually include surveillance culture, contact tracing, isolation of carriers and environmental disinfection. Nevertheless, isolation facilities are not always readily available, particularly in resource-limited regions. In addition, contact isolation may result in various adverse effects on the mental well-being of isolated patients, such as depression, anxiety and anger. Time spent with patients in isolation by healthcare workers is less, with a negative effect on patient safety with an eight-fold increase in the risk of adverse events due to supportive care failure.

There has been a growing interest in extending FMT for the decolonization of CRE. However, most of the studies are limited to case reports or case series with small sample sizes (ranging from 10 to 39 patients) as shown by a recent systematic review. The pooled rate of CRE decolonization is promising at 62.1%. However, a randomized controlled trial (RCT) remains the most optimal study design to investigate the true beneficial effect of FMT on CRE decolonization. FMT via enema route has several advantages over upper GI delivery or colonoscopy. First, the administration of fecal suspension via a feeding tube may not be acceptable to some patients. Second, colonoscopy carries complications of gut perforation, aspiration, and cardiopulmonary suppression from the use of sedatives, in particular among frail and elder patients.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged 18 or above admitted to the medical ward of Queen Mary Hospital, the teaching hospital of the University of Hong Kong
* Rectal swabs or stool specimens showing the presence of CRE
* Positive CRE specimen within one week of commencement

Exclusion Criteria:

* Pregnancy
* Severe immunodeficiency (e.g. advanced human immunodeficiency virus infection (CD4 lymphocyte count ≤200/mm3), myelosuppressive chemotherapy)
* Significant neutropenia (absolute neutrophil count ≤1.0 x 109/L)
* Recent antibiotic use within 30 days prior to consent
* Contraindications for retention enema (intestinal obstruction, ileus and gut perforation).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-08-19 (Estimated); Study Completion 2025-08-19 (Estimated)

PRIMARY OUTCOMES:
CRE clearance rate | 1 month post-FMT
  CRE clearance rate via enema

SECONDARY OUTCOMES:
CRE clearance rate | 1 week, 2 week, 3 month, 6 month and 12 month post-FMT
  CRE clearance rate post-FMT
All-cause mortality | 1 month, 3 month, 6 month and 12 month post-FMT
  All-cause mortality post-FMT

CONTACTS AND LOCATIONS:
Overall Officials: Ka Shing Cheung, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Backman C, Taylor G, Sales A, Marck PB. An integrative review of infection prevention and control programs for multidrug-resistant organisms in acute care hospitals: a socio-ecological perspective. Am J Infect Control. 2011 Jun;39(5):368-378. doi: 10.1016/j.ajic.2010.07.017. Epub 2011 Mar 23. PMID 21429622
- [Background] Quraishi MN, Widlak M, Bhala N, Moore D, Price M, Sharma N, Iqbal TH. Systematic review with meta-analysis: the efficacy of faecal microbiota transplantation for the treatment of recurrent and refractory Clostridium difficile infection. Aliment Pharmacol Ther. 2017 Sep;46(5):479-493. doi: 10.1111/apt.14201. Epub 2017 Jul 14. PMID 28707337
- [Background] Macareno-Castro J, Solano-Salazar A, Dong LT, Mohiuddin M, Espinoza JL. Fecal microbiota transplantation for Carbapenem-Resistant Enterobacteriaceae: A systematic review. J Infect. 2022 Jun;84(6):749-759. doi: 10.1016/j.jinf.2022.04.028. Epub 2022 Apr 21. PMID 35461908